CLINICAL TRIAL: NCT04694365
Title: A Open, Single-dose, Parallel-control Study to Investigate the Pharmacokinetics of Fluzoparib in Healthy Subjects and Those With Impaired Liver Function.
Brief Title: Safety and Pharmacokinetics of Fluzoparib in Healthy Subjects and Those With Impaired Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SHR3162-I-117
Record Dates: First submitted 2020-12-28; First posted 2021-01-05 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Hepatic Impairment; Healthy Subjects
MeSH Terms: interventions — fluzoparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal Hepatic Function (Experimental)
  Interventions: Drug: Fluzoparib
- Mild Hepatic Impairment (Experimental)
  Interventions: Drug: Fluzoparib
- Moderate Hepatic Impairment (Experimental)
  Interventions: Drug: Fluzoparib

INTERVENTIONS:
Drug: Fluzoparib — A single oral dose of 50 mg Fluzoparib will be administered.

SUMMARY:
This study is designed to evaluate the safety and pharmacokinetics of Fluzoparib in subjects with impaired liver function in comparison with healthy subjects ,to develop dose recommendations for patients with hepatic impairment.

ELIGIBILITY:
Inclusion Criteria for subjects with impaired liver function:

1. Sign the informed consent before the trial, and fully understand the trial content, process and possible adverse reactions;
2. Ability to complete the study as required by the protocol;
3. Healthy male or female subjects aged 18 to 65 (including 18 and 45) at the date of signing the informed consent;
4. Male body weight ≥ 50 kg, female body weight ≥ 45 kg, and body mass index (BMI) within the range of 19 ~ 29kg /m2 (including 19 and 29);
5. Participants with alcoholic liver disease, autoimmune liver disease, Non-Alcoholic Liver Diseases and inherited metabolic liver disease. Mild Hepatic Impairment group should be stable≥28days ; Moderate Hepatic Impairment group should be stable≥14days.

Exclusion Criteria impaired liver function:

1. Allergic constitution;
2. History of drug use, or drug abuse screening positive;
3. Alcoholic or often drinkers;
4. Received any surgery in the previous 6 months before screen phase;
5. A clear medical history of important primary organ diseases such as nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolism and musculoskeletal sysem.
6. Abnormal clinical laboratory tests and clinical significance judged by the investigator or other clinical findings showing the following diseases, including but not limited to gastrointestinal tract, kidney, liver, nerve, blood, endocrine, tumor, lung, immune, mental or cardiovascular and cerebrovascular diseases.
7. Patients with hepatic encephalopathy;
8. Taking any drugs which affects the metabolic enzyme CYP3A within 14 days before the study started,

Inclusion Criteria for subjects with normal liver function:

1. Sign the informed consent before the trial, and fully understand the trial content, process and possible adverse reactions;
2. Ability to complete the study as required by the protocol;
3. Healthy male or female subjects aged 18 to 65 (including 18 and 45) at the date of signing the informed consent;The age and gender should match with impaired liver function;
4. Male body weight ≥ 50 kg, female body weight ≥ 45 kg, and body mass index (BMI) within the range of 19 ~ 29kg /m2 (including 19 and 29); The body weight should match with impaired liver function.

Exclusion Criteria normal liver function:

1. Allergic constitution;
2. History of drug use, or drug abuse screening positive;
3. Alcoholic or often drinkers;
4. Received any surgery in the previous 6 months before screen phase;
5. A clear medical history of important primary organ diseases such as nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolism and musculoskeletal sysem.
6. Abnormal clinical laboratory tests and clinical significance judged by the investigator or other clinical findings showing the following diseases, including but not limited to gastrointestinal tract, kidney, liver, nerve, blood, endocrine, tumor, lung, immune, mental or cardiovascular and cerebrovascular diseases.
7. Taking any drugs which affects the metabolic enzyme CYP3A within 14 days before the study started,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameters of Fluzoparib: Cmax | through study completion, an averange of half year
Pharmacokinetics parameters of Fluzoparib: AUC0-t | through study completion, an averange of half year
Pharmacokinetics parameters of Fluzoparib: AUC0-∞(if available) | through study completion, an averange of half year

SECONDARY OUTCOMES:
Other pharmacokinetics parameters of Fluzoparib: Tmax | through study completion, an averange of half year
plasma protein binding rate of Fluzoparib | through study completion, an averange of half year
The incidence and severity of adverse events/serious adverse events (based on NCI-CTCAE 5.0) | through study completion, an averange of half year
Other pharmacokinetics parameters of Fluzoparib: T1/2 etc. | through study completion, an averange of half year

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Infectious Diseases Hospital, Zhengzhou, Henan, China